CLINICAL TRIAL: NCT06197659
Title: The Effect of Peroperative Restrictive and Liberal Fluid Regimens on Postoperative Nausea-vomiting and Quality of Recovery in Laparoscopic Cholecystectomy: a Prospective Randomized Study.
Brief Title: Effect of Liberal and Restrictive Fluids on Nausea-vomiting
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karaman Training and Research Hospital (Other)
Responsible Party: Principal Investigator, muhammet korkusuz, Principal Investigator, MD, Karaman Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 10-2023/14
Record Dates: First submitted 2023-12-12; First posted 2024-01-09 (Actual); Last update posted 2024-02-16 (Actual); Status verified 2024-02

CONDITIONS: Postoperative Nausea and Vomiting
Keywords: Postoperative Nausea and Vomiting; Laparoscopic Cholecystectomy
MeSH Terms: conditions — Postoperative Nausea and Vomiting

STUDY DESIGN:
Intervention Model Description: There are two group;
  1. Experimental Group: Group L; Liberal Fluid Group; Peroperative 20 mL/kg/h intravenous ringer lactate will be administered.
  2. Sham Comparator: Group R; Restrictive Fluid Group; Peroperative 5 mL/kg/h intravenous ringer lactate will be administered.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: patients, care providers, and outcome assessors will be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Liberal Fluid Group (Active Comparator): Patients in this group will be administered 20 mL/kg/h ringer lactate intravenously peroperatively.
  Interventions: Other: Liberal Fluid Grubu
- Restrictive Fluid Group (Sham Comparator): Patients in this group will be administered 4 mL/kg/h ringer lactate intravenously peroperatively.
  Interventions: Other: Restrictive Fluid Group

INTERVENTIONS:
Other: Liberal Fluid Grubu — Patients in this group will be administered 20 mL/kg/h ringer lactate intravenously peroperatively.
  Other Names: Liberal group
  Arms: Liberal Fluid Group
Other: Restrictive Fluid Group — Patients in this group will be administered 4 mL/kg/h ringer lactate intravenously peroperatively.
  Other Names: Restrictive group
  Arms: Restrictive Fluid Group

SUMMARY:
Patients planned for laparoscopic cholecystectomy will be included in this study. The effects of liberal and restrictive fluid regimens given peroperatively to patients undergoing laparoscopic cholecystectomy will be compared on postoperative nausea and vomiting. The aim of this study is to investigate which regimen is more effective on postoperative nausea and vomiting in laparoscopic cholecystectomy.

DETAILED DESCRIPTION:
Postoperative nausea and vomiting (PONV) is a common and disturbing side effect of anesthesia and surgery, and while its incidence in all surgical procedures varies between 20-77% if antiemetic prophylaxis is not applied, this rate is even higher in people prone to vomiting, such as cyclic vomiting syndrome . Its incidence varies between 53 - 72%, especially in patients undergoing laparoscopic cholecystectomy surgery, if antiemetic prophylaxis is not administered.

Since most existing antiemetics are expensive and cannot completely eliminate PONV, pharmacological PONV prophylaxis may not be cost-effective. For this reason, the incidence of PONV can be reduced by increasing the amount of inexpensive fluid used during surgery instead of prophylactic drug treatment. There are several studies investigating the effect of different perioperative fluid administration schemes on PONV in the adult population, especially in patients undergoing laparoscopic cholecystectomy or gynecological surgery, with variable results.

Based on this point, the inestigetors wanted to examine the effect of perioperative liberal and restrictive fluid treatments on PONV in patients who underwent laparoscopic cholecystectomy.

ELIGIBILITY:
Inclusion Criteria:

* Patients planned for laparoscopic cholecystectomy
* Patients aged 18-70

Exclusion Criteria:

* Congestive heart failure.
* Diabetes.
* Epilepsy.
* Heart valve disease.
* They are pregnant.
* Chronic liver disease.
* Chronic kidney disease. Chronic gastrointestinal tract disease. Those who used antiemetic drugs within 24 hours before surgery. Those who developed intraoperative hypertension. Those who develop excessive blood loss. Patients whose surgery procedure takes more than 2 hours.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-02-10 (Actual); Study Completion 2024-02-15 (Actual)

PRIMARY OUTCOMES:
Incidence of postoperative nausea-vomiting | Postoperative 24 hours
  Incidence of nausea and vomiting within 24 hours after surgery. The presence of at least one episode of nausea, retching and vomiting in the first 24 hours postoperatively will be considered a positive result.
Quality of recovery | Postoperative 24 hours
  Quality of recovery will be evaluated at the 24th hour using the QoR-15 scale. It is a scale consisting of 15 questions and scoring from 0 to 10 for each question. 0 represents the worst and 150 represents the best recovery quality.

SECONDARY OUTCOMES:
Time to first antiemetic request | Postoperative 24 hours
  Time to first antiemetic request within 24 hours after surgery
Time to request first oral drink | Postoperative 24 hours
  Time to request first oral drink within 24 hours after surgery
First mobilization time | Postoperative 24 hours
  First mobilization time after surgery
Total amount of analgesic | Postoperative 24 hours
  Total amount of rescue analgesic (tramadol) in the 24 hours after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Muhammet Korkusuz, Principal Investigator — Karamanoglu Mehmetbey University, School of Medicine
Locations (1):
- Karaman Taining and Research Hospital, Karaman, Turkey (Türkiye)